CLINICAL TRIAL: NCT06961903
Title: Comparison of the Effectiveness of Functional Taping, Manual Therapy and Stereodynamic Interference Current in Patients With Chronic Low Back Pain
Brief Title: Effectiveness of Functional Taping, Manual Therapy and Stereodynamic Interference Current
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Collaborators: Acibadem Atakent University Hospital (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Muhammed Fatih Kavak, Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/15
Record Dates: First submitted 2025-04-29; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Chronic Low Back Pain (Non-specific, Uncomplicated)
Keywords: Chronic low back pain; manual therapy; functional taping; electrotherapy; kinesiophobia
MeSH Terms: conditions — Kinesiophobia | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant
Masking Description: This study was conducted with single-blind masking, where the participants were blinded to the group allocation. Participants were not informed about the specific physiotherapy technique or intervention they received (e.g., whether they received functional taping, manual therapy, or stereodynamic interference current) to minimize expectation bias. However, due to the nature of the interventions, therapists administering the treatment were not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- physiotherapy (Experimental): A program consisting of therapeutic ultrasound, hot pack, massage, and McKenzie exercises was administered as the intervention.
  Interventions: Other: physiotherapy programme
- Functional Taping (Experimental): A program consisting of therapeutic ultrasound, hot pack, massage, and McKenzie exercises was administered as the intervention. In addition, the taping method applied in this study can be defined as a "Function-Oriented Taping Application to Preserve Extension: Lumbar Extension Taping," which was specifically designed to maintain lumbar extension.
  Interventions: Other: physiotherapy programme; Other: Functional Taping
- Manual Therapy (Experimental): A program consisting of therapeutic ultrasound, hot pack, massage, and McKenzie exercises was administered as the intervention.Manual Therapy (MT), which literally means "hands-on treatment," is an evidence-based therapeutic approach consisting of skilled hand movements and maneuvers applied to produce therapeutic effects and to treat musculoskeletal dysfunctions and pain. In addition to the standard program, manual therapy was also administered in this study.
  Interventions: Other: physiotherapy programme; Other: Manual Therapy
- Stereodynamic Interference Current (Experimental): A program consisting of therapeutic ultrasound, hot pack, massage, and McKenzie exercises was administered as the intervention.In addition, the stereodynamic interference current method was applied in this study. A 'Y' electrode was used during the application. Due to the rapid development of accommodation, the current intensity was frequently increased during the session. The average treatment duration was 15 minutes, and a frequency of 50-100 Hz was used to achieve analgesic effects.
  Interventions: Other: physiotherapy programme; Other: Stereodynamic Interference Current

INTERVENTIONS:
Other: physiotherapy programme — A program consisting of therapeutic ultrasound, hot pack, massage, and McKenzie exercises was administered as the intervention.
Other: Functional Taping — A program consisting of therapeutic ultrasound, hot pack, massage, and McKenzie exercises was administered as the intervention. In addition, the taping method applied in this study can be defined as a "Function-Oriented Taping Application to Preserve Extension: Lumbar Extension Taping," which was specifically designed to maintain lumbar extension.
  Arms: Functional Taping
Other: Manual Therapy — A program consisting of therapeutic ultrasound, hot pack, massage, and McKenzie exercises was administered as the intervention.Manual Therapy (MT), which literally means "hands-on treatment," is an evidence-based therapeutic approach consisting of skilled hand movements and maneuvers applied to produce therapeutic effects and to treat musculoskeletal dysfunctions and pain. In addition to the standard program, manual therapy was also administered in this study.
  Arms: Manual Therapy
Other: Stereodynamic Interference Current — A program consisting of therapeutic ultrasound, hot pack, massage, and McKenzie exercises was administered as the intervention.In addition, the stereodynamic interference current method was applied in this study. A 'Y' electrode was used during the application. Due to the rapid development of accommodation, the current intensity was frequently increased during the session. The average treatment duration was 15 minutes, and a frequency of 50-100 Hz was used to achieve analgesic effects.
  Arms: Stereodynamic Interference Current

SUMMARY:
This study aimed to compare the effects of functional taping, manual therapy, and stereodynamic interference current applications on pain, functional capacity, sleep quality, and kinesiophobia in individuals with chronic low back pain (LBP). Conducted with 88 participants, the study divided them into four groups: a control group (standard physiotherapy), a functional taping group, a manual therapy group, and a stereodynamic interference current group. All groups received 10 sessions of treatment, 3 days a week. The study evaluated pain intensity (VAS), fear of movement (FOM), functional disability (ODI), and sleep quality (PSQI) at three points: before treatment, after treatment, and one month later. Results showed that manual therapy significantly improved pain levels (p<0.05), while stereodynamic interference current also reduced pain. Functional taping was most effective in reducing kinesiophobia (p<0.05). No significant differences were observed between the groups in terms of the Oswestry Disability Index and Pittsburgh Sleep Quality Index scores (p>0.05). The study concluded that manual therapy was the most effective for pain control, and functional taping was superior for managing kinesiophobia, emphasizing the need for individualized and multidisciplinary approaches in treating musculoskeletal health issues.

DETAILED DESCRIPTION:
This randomized controlled experimental study was designed to compare the effects of functional taping, manual therapy, and stereodynamic interference current applications on pain, functional capacity, sleep quality, and kinesiophobia in individuals with chronic low back pain (LBP). A total of 88 participants diagnosed with chronic LBP were recruited and randomly assigned into four groups: a control group receiving standard physiotherapy, a functional taping group, a manual therapy group, and a stereodynamic interference current group.

All participants underwent treatment for 10 sessions, administered three times per week. The interventions were standardized across the groups, and treatment adherence was carefully monitored. Assessments were conducted at three time points: baseline (before treatment), immediately after the treatment period, and one month following the completion of treatment.

The primary outcome measures included pain intensity, assessed with the Visual Analog Scale (VAS); fear of movement (kinesiophobia), assessed with the Tampa Scale of Kinesiophobia (TSK); functional disability, assessed with the Oswestry Disability Index (ODI); and sleep quality, assessed with the Pittsburgh Sleep Quality Index (PSQI).

The results indicated that the manual therapy group exhibited the greatest improvement in both resting and movement-related pain (p<0.05). Stereodynamic interference current application was also found to significantly reduce pain levels. The functional taping group demonstrated the most substantial improvement in reducing kinesiophobia scores (p<0.05). However, there were no statistically significant differences between the groups regarding functional disability (ODI) and sleep quality (PSQI) scores (p>0.05).

The findings highlight that manual therapy is particularly effective for managing pain in chronic LBP patients, while functional taping is especially beneficial for addressing fear of movement. These results underscore the importance of individualized treatment planning based on the specific needs of patients and support the integration of multidisciplinary approaches to effectively manage complex musculoskeletal conditions

ELIGIBILITY:
Inclusion Criteria:

* participants had to be aged between 20 and 50 years,
* have a diagnosis of chronic low back pain (low back pain persisting for more than 12 weeks),
* have a Visual Analogue Scale (VAS) score of at least 4/10,
* be suitable for physical therapy, and sign a written informed consent form by voluntarily agreeing to participate in the study.

Exclusion Criteria:

* with a history of lumbar surgery,
* acute inflammatory diseases or signs of infection, rheumatological, neurological or cardiovascular system diseases,
* pregnancy status,
* history of invasive intervention in the lumbar region within the last six months

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
pain intensity | through study completion, an average of one month.
  The VAS is a measurement tool that allows individuals to subjectively assess the intensity of pain they perceive. The VAS is usually located on a 10 cm long horizontal line between two extremes ranging from 'no pain' to 'unbearable pain'. Participants are asked to mark their current pain level on this line and the measurement is made by evaluating the distance from the marked point to the starting point in centimetres (cm). The VAS is a simple and reliable tool that is frequently preferred to quantitatively measure the severity of pain, especially in clinical research.
kinesiophobia level | through study completion, an average of one month.
  The Tampa Kinesiophobia Scale (TSK) is a self-report form developed to measure the fear of movement that individuals develop due to pain. The TSK consists of a total of 17 items and each item is scored from 'strongly disagree' to 'strongly agree' on a 4-point Likert-type scale. High scores indicate a high level of movement avoidance and pain-related fear of movement. Especially in individuals with chronic pain, it is an important tool in terms of evaluating the fear of movement related to pain and making plans for treatment.
Low Back Disability Index | through study completion, an average of one month.
  The Oswestry Low Back Disability Index (ODI) is a comprehensive scale developed to assess the level of functional disability in individuals with low back pain and measures the impact of low back pain on activities of daily living. This index, which consists of a total of 10 items, evaluates daily activities such as pain intensity, personal care, lifting, walking, sitting, sitting, standing, sleeping, social life, travelling and sex life. Each item is scored between 0 and 5 and the level of disability is determined by converting the total score into a percentage. Higher scores mean more disability. The ODI is one of the most widely used tools worldwide to measure functional status in individuals with chronic low back pain.
Sleep Quality Index | through study completion, an average of one month.
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report scale developed to assess the sleep quality of individuals in the last month. The PSQI consists of a total of 19 items and assesses seven different components, including sleep duration, sleep latency, sleep efficiency, sleep disturbances, sleep medication use, and daytime sleepiness. The scores obtained from each component are included in the total scoring to determine the overall sleep quality. The total score obtained varies between 0 and 21; high scores indicate poor sleep quality. PSQI is a reliable measurement tool to detect sleep quality deterioration especially in chronic pain patients.

CONTACTS AND LOCATIONS:
Locations (1):
- acibadem Hospital, Istanbul, Turkey (Türkiye)